CLINICAL TRIAL: NCT03334929
Title: Virtual Reality Distraction for Anxiety Reduction During Trigger Points Procedures in Pain Medicine Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1088873
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Pain Management
Keywords: virtual reality; trigger point injections
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality intervention (Experimental): Participants will be wearing Virtual Reality headset called Oculus gear equipped with Samsung galaxy S7 during the trigger point injections. The VR app chosen is called Relax VR - Rest, Relaxation & Meditation, which will provide a calm beach scene with waves and soothing musics.
  Interventions: Device: Virtual Reality headset
- control (No Intervention): Participants in this group will receive trigger point injections without any intervention. The trigger point injections will be performed in daily manner.

INTERVENTIONS:
Device: Virtual Reality headset — The participants in this group would wear Virtual Reality headset called Oculus Gear VR during their trigger point injections.
  Arms: Virtual Reality intervention

SUMMARY:
This study aims to evaluate the effect of Virtual Reality (VR) as a distraction method to help those patients undergoing trigger points therapy to reduce anxiety and increase patient satisfaction. Half of the participants will wear VR gear, meanwhile the other half will be in control group, which will not wear VR headset, only the normal care.

DETAILED DESCRIPTION:
trigger points can cause a wide range of pain symptoms; pain in the anterior shoulder and down the arm, headache pain, back pain, hip pain, knee pain, frozen shoulder pain, and other symptoms. Local anesthetic injections and lidocaine injections are common "wet" needling treatments for trigger points injections. The proposed mechanism by which trigger points injections alleviate pain is based on mechanical disruption of the taut bands of muscle with palpation based needling. During injections, patients may feel an intensified pain and a twitch response.

Distraction has been proved to be an effective tool in pain management, and it can also be used for a variety of medical procedures. By engaging in assigned tasks, pain and anxiety are assumed to be lessened throughout the procedure, while leaving patients less occupied by pain stimuli. . An immersive virtual environment may be preferable to medications such as sedatives, due to side effects and prolonged discharge from procedure suite. Occasionally, medications may not even be available in a busy interventional pain suite. At the UCD pain clinic, we do not offer sedating medications for bedside procedures like trigger point injections. By wearing VR headset, patients may feel less tense, anxious, and painful during trigger point injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old, who are referred to UC Davis Pain Medicine Clinic and are candidates for trigger point injections, are English speaking and can understand oral and written instructions

Exclusion Criteria:

* Patients who have high risk of motion sickness, seizure disorder, visual/hearing impairment, prisoners or are pregnant are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level | Immediately pre- and post-procedure
  Spielberger State-Trait Anxiety Inventory items measuring state anxiety. All items are rated on a 4-point scale, with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Change in pain score | Immediately pre- and post-procedure
  Participants will be asked to indicate pain score in a scale of 0-10, with higher scores indicating greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Naileshni Singh, MD, Principal Investigator — University of California, Davis; Samir Sheth, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerwin RD. Myofascial Trigger Point Pain Syndromes. Semin Neurol. 2016 Oct;36(5):469-473. doi: 10.1055/s-0036-1586262. Epub 2016 Sep 23. PMID 27704503
- [Background] Zhou JY, Wang D. An update on botulinum toxin A injections of trigger points for myofascial pain. Curr Pain Headache Rep. 2014 Jan;18(1):386. doi: 10.1007/s11916-013-0386-z. PMID 24338700
- [Background] Scott NA, Guo B, Barton PM, Gerwin RD. Trigger point injections for chronic non-malignant musculoskeletal pain: a systematic review. Pain Med. 2009 Jan;10(1):54-69. doi: 10.1111/j.1526-4637.2008.00526.x. Epub 2008 Nov 5. PMID 18992040
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326